CLINICAL TRIAL: NCT02319564
Title: Randomized Trial Assessing the Effectiveness of Beclomethasone and Combination Beclomethasone and Salbutamol as Compared With Placebo in Preschool Aged Children With Wheeze
Brief Title: Combined Glucocorticoid Adrenergic Therapy For Wheezy Preschool Children
Acronym: CONjuGATE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study population too narrow - unable to recruit any patients.
Sponsor: University of Calgary (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, David W Johnson, Professor, Departments of Pediatrics, Pharmacology & Physiology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ConRCT1
Record Dates: First submitted 2014-11-30; First posted 2014-12-18 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Wheeze
Keywords: Wheeze; Asthma; Randomized Trial; Pre-school aged children
MeSH Terms: conditions — Respiratory Sounds; Asthma | interventions — Beclomethasone; Albuterol; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- beclomethasone (Active Comparator): beclomethasone dipropionate 250mcg per puff per puff (Chiesi metered dose inhaler) via a masked spacer (Aerochamber Max®, Plattsburgh, NY, USA). One puff BID for 14 days.
  Non-identifiable MDI prepared by Chiesi Farmaceutici Inc.
  Interventions: Drug: Beclomethasone; Device: Aerochamber Max®
- beclomethasone and salbutamol (Active Comparator): beclomethasone diprionate 250mcg and salbutamol 100mcg per puff (Chiesi metered dose inhaler) via a masked spacer (Aerochamber Max®, Plattsburgh, NY, USA). One puff BID for 14 days.
  Non-identifiable MDI prepared by Chiesi Farmaceutici Inc.
  Interventions: Drug: Beclomethasone and Salbutamol; Device: Aerochamber Max®
- Placebo (Placebo Comparator): placebo (Chiesi metered dose inhaler) via a masked spacer (Aerochamber Max®, Plattsburgh, NY, USA). One puff BID for 14 days.
  Non-identifiable MDI prepared by Chiesi Farmaceutici Inc.
  Interventions: Drug: Placebo; Device: Aerochamber Max®

INTERVENTIONS:
Drug: Beclomethasone
  Other Names: Clenil
  Arms: beclomethasone
Drug: Beclomethasone and Salbutamol
  Other Names: Clenil Compositum
  Arms: beclomethasone and salbutamol
Drug: Placebo
  Arms: Placebo
Device: Aerochamber Max®
  Other Names: Masked Spacer for metered dose inhaler

SUMMARY:
The investigators goal is to conduct a pilot randomized controlled trial (RCT) whose purpose is to determine the feasibility of a randomized trial designed to determine if either inhaled beclomethasone or a combination of inhaled beclomethasone/salbutamol (Clenil Compositum) are superior to placebo in treating pre-school aged children with an acute wheezing episode.

ELIGIBILITY:
Inclusion Criteria:

1. children 12-60 months of age
2. wheeze on auscultation
3. mild respiratory distress as measured by a score of < 3 on the Pediatric Respiratory Assessment Measure (PRAM)
4. discharged home after evaluation by their ED physician.

Exclusion Criteria:

1. treatment with oral or parenteral corticosteroids in the last 14 days
2. treatment with more than 2 doses of inhaled corticosteroids in the previous seven days
3. presence of a severe co-morbidity such as bronchopulmonary dysplasia, cystic fibrosis, congenital heart disease, adrenal disorder or immune deficiency
4. previously enrolled into this study or concurrently enrolled in another intervention trial
5. lack of telephone access or presence of a significant language barrier

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduce unplanned-symptomatic visits to clinicians | After enrolment is complete

SECONDARY OUTCOMES:
Reduce the number of days with respiratory symptoms | Will be analyzed 1-2 months after enrolment is complete, looking at the full follow-up period of 21 days
Reduce the need for rescue salbutamol use | Will be analyzed 1-2 months after enrolment is complete, looking at the full follow-up period of 21 days
Reduce hospitalization rates of target population | Will be analyzed 1-2 months after enrolment is complete, looking at the full follow-up period of 21 days
Reduce overall societal health care costs of target population | Will be analyzed 1-2 months after enrolment is complete, looking at the full follow-up period of 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No